CLINICAL TRIAL: NCT00182650
Title: Pilot/Feasibility Study To Evaluate The Safety Of Cellular Immunotherapy For CD19+ Follicular Lymphoma Using Autologous Cytolytic T Cells Genetically-Modified To Be CD19-Specific And Co-Express HyTK
Brief Title: Cellular Adoptive Immunotherapy in Treating Patients With Relapsed or Refractory Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000438797; R21CA105824 (NIH); P30CA033572 (NIH); CHNMC-IRB-01160
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — aldesleukin; Rituximab; fludarabine phosphate

INTERVENTIONS:
Biological: aldesleukin
Biological: rituximab
Biological: therapeutic autologous lymphocytes
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Cellular adoptive immunotherapy uses a person's white blood cells that are treated in the laboratory to stimulate the immune system in different ways and stop cancer cells from growing. Rituximab and fludarabine may also prevent the body from making an immune response against the laboratory-treated white blood cells that are put back into the body. Interleukin-2 may help the laboratory-treated white blood cells stay in the body longer. Giving cellular adoptive immunotherapy together with rituximab, fludarabine, and interleukin-2 may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects of cellular adoptive immunotherapy in treating patients with relapsed or refractory follicular non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of cellular adoptive immunotherapy using autologous cytotoxic T lymphocytes genetically modified to express a CD19-specific chimeric immunoreceptor gene and HyTK selection/suicide gene in patients with relapsed or refractory follicular non-Hodgkin's lymphoma.

Secondary

* Determine the in vivo persistence of adoptively transferred cytolytic T cells in patients treated with lymphodepleting therapy comprising rituximab and fludarabine.
* Assess the development of host immune responses against the CD19-specific chimeric immunoreceptor gene and/or HyTK selection/suicide gene.
* Determine the safety of low-dose interleukin-2 in supporting in vivo persistence of adoptively transferred cytotoxic T cells.
* Determine the anti-tumor activity of this regimen in these patients.

OUTLINE: This is a nonrandomized, open-label, pilot study.

* Leukapheresis: Patients undergo leukapheresis for collection of peripheral blood mononuclear cells (PBMCs). CD3-positive cytotoxic T lymphocytes (CTLs) are isolated and genetically modified to express a CD19-specific chimeric immunoreceptor and the HyTK fusion protein, and are then expanded in vitro.
* Lymphodepleting therapy: Patients receive rituximab and fludarabine prior to T-cell infusions.
* Cellular adoptive immunotherapy and interleukin-2 (IL-2): Patients receive a total of 5 infusions of genetically modified autologous T cells. Patients may receive low-dose IL-2 subcutaneously after infusions 3, 4, and 5.
* Additional IL-2 therapy: After the completion of the last T-cell infusion, patients with evidence of adoptively transferred T cells may receive additional IL-2.

After completion of study treatment, patients are followed periodically for approximately 65 days and then annually for at least 15 years.

PROJECTED ACCRUAL: At least 5 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular non-Hodgkin's lymphoma (NHL)

  * High-risk disease, as defined by any of the following:

    * Relapsed within 6 months after the last treatment
    * Failed to achieve a complete response during the last treatment
    * Relapsed after prior autologous hematopoietic stem cell transplantation (HSCT)
* No current transformation of lymphoma (e.g., elements of intermediate- or high-grade lymphoma by biopsy)
* No active CNS disease by lumbar puncture or radiology scan NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 16 to 70

Performance status

* Karnofsky 50-100%

Life expectancy

* More than 16 weeks

Hematopoietic

* Absolute neutrophil count > 500/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)* (unless due to Gilbert's disease)
* ALT ≤ 2.5 times ULN* NOTE: *Unless due to NHL

Renal

* Creatinine ≤ 1.5 times ULN* OR
* Creatinine clearance ≥ 80 mL/min* NOTE: *Unless due to NHL

Immunologic

* HIV negative
* Epstein-Barr virus positive
* No history of allergy or intolerance to ganciclovir

Other

* Negative pregnancy test
* No history of another malignancy except basal cell skin cancer or carcinoma in situ
* No other uncontrolled or severe illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior allogeneic HSCT
* No other immunotherapy during and for approximately 65 days after the last T-cell infusion, unless approved by the Principal Investigator (PI)

Chemotherapy

* No other chemotherapy during and for approximately 65 days after the last T-cell infusion, unless approved by the PI

  * Patients may receive chemotherapy after leukapheresis while waiting for CD19-specific T cells to be manufactured

Endocrine therapy

* No systemic corticosteroids during and for approximately 65 days after the last T-cell infusion, unless approved by the PI

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent participation in another investigational study
* No immunosuppression agents or other investigational agents during and for approximately 65 days after the last T-cell infusion, unless approved by the PI

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2004-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States